CLINICAL TRIAL: NCT05386342
Title: A Post-market Clinical Study to Confirm the Performance and Safety of the LeMaitre TufTex Over-the-Wire (OTW) Embolectomy Catheter on Patients Undergoing Surgical Treatment for the Removal of Arterial Emboli and/or Thrombi
Brief Title: A PMCF Study Confirm the Performance and Safety of the TufTex Over-the-Wire (OTW) Embolectomy Catheters
Acronym: OTW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LeMaitre Vascular (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-16-002
Record Dates: First submitted 2022-05-10; First posted 2022-05-23 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Thrombus; Embolus; Occlusion; Vessel
MeSH Terms: conditions — Thrombosis; Embolism; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- LeMaitre TufTex Over-the-Wire Embolectomy Catheter (Other): The LeMaitre Over the Wire Embolectomy Catherer is indicated for use in the removal of emboli and thrombi during embolectomy and/or thrombectomy. It can also be used for catheter placement over a guidewire, vessel occlusion, fluid infusion and/or aspiration.
  Interventions: Device: TufTex Over-the-Wire Embolectomy Catheter

INTERVENTIONS:
Device: TufTex Over-the-Wire Embolectomy Catheter — The OTW Catheter can be used for the removal of emboli and thrombi. It can also be used for catheter placement over a guidewire, vessel occlusion, fluid infusion and/or aspiration.

SUMMARY:
A PMCF study to confirm the performance and safety of the LeMaitre® TufTex Over-the-Wire Embolectomy Catheter

DETAILED DESCRIPTION:
This clinical investigation is a prospective, single-arm, multicenter, post-market study to proactively collect clinical data on the LeMaitre® TufTex Over-the-Wire (OTW) Embolectomy Catheters and to confirm its performance in removing arterial emboli and/or thrombi, to identify and analyze emergent risks on the basis of factual evidence, and to ensure the continued acceptability of the benefit/risk ratio. The intended purpose of the device in this post market clinical study is identical to the indication of use of the device.

The TufTex OTW post-market study is initiated by the Sponsor and manufacturer of the device, LeMaitre Vascular, Inc.

The investigation will take place in 4 sites, most likely in 3 different countries. A total number of 112 subjects is anticipated to be enrolled, who are intended to undergo surgical treatment for the removal of a emboli and/or thrombi. The anticipated enrollment period is 48 months, and the participation per subject is 1 month. The total study duration is expected to be 56 months (4 months start-up, 48 months of recruitment, 1 month of follow-up, 3 months of closure.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subject, ≥ 18 years of age at time of enrollment.
2. Subject who is scheduled to undergo surgical treatment for the removal of an emboli or thrombi during an embolectomy and/or thrombectomy procedure, where one of the LeMaitre® Embolectomy Catheter will be used.
3. Subject signed an Informed Consent for participation.
4. Subject diagnosed with a embolus/thrombus.
5. Subjects for whom thrombolytic therapy had failed or was contraindicated.

Exclusion Criteria:

1. Co-morbidity that in the discretion of the investigator might confound the results.
2. Subjects who are unable to read or write.
3. Pregnant or lactating women at time of enrollment
4. Subjects who are immune compromised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Performance objective is the technical success being <30% residual stenosis | 1 month post index procedure
  The primary performance objective of the study is the technical success as defined as <30% residual stenosis of the target vessel as evaluated on the completion digital subtraction angiography (DSA).
Safety objective is defined as acceptable safety outcomes during the procedure and at follow-up | 1 month post index procedure
  The primary safety objective is defined as acceptable safety outcomes (e.g. (Serious) Device and/or Procedure Related Events) during the procedure and 1 Month post index procedure.

SECONDARY OUTCOMES:
1.Clinical success | 1 month post index procedure
  Clinical success is target vessel dependent and defined as; 1. the absence of target vessel limb amputation post-intervention in case of limb cloths, and 2. successful dialysis sessions performed post-intervention in case of dialysis shunt revascularization
2. Revision rate | 1 month post index procedure
  Revision rate is defined as the number of patients with target vessel reintervention
3. Primary assisted patency | 1 month post index procedure
  Primary assisted patency is defined as target vessel patency; the target vessel is patent but there may have been some intervention required to maintain that patency.
4. Secondary patency | 1 month post index procedure
  Secondary patency is defined as the target vessel patency including target vessel that have been occluded and there has been an intervention to restore patency

OTHER OUTCOMES:
Exploratory endpoints | 1 month post index procedure
  Number of LeMaitre® TufTex OTW Embolectomy Catheters used per intervention

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Prouse, MD, Principal Investigator — Ospedale Regionale di Lugano - sede Civico; Andrej Udelnow, MD, Principal Investigator — University of Brandenburg; Sandra Korn, MD, Principal Investigator — University Hospital Carl Gustav Carus
Locations (3):
- Germany (2):
  - Andrej Udelnow, Brandenburg
  - University Hospital Carl Gustav Carus TU Dresden, Dresden
- Ospedale Regionale di Lugano - sede Civico, Lugano, Switzerland